CLINICAL TRIAL: NCT05007145
Title: A Randomized, Open-label, Phase II Study of PD-1 Inhibitor Combined With Neoadjuvant Chemotherapy Versus Neoadjuvant Chemoradiotherapy in Subjects With Resectable Locally Advanced Thoracic Esophageal Squamous Cell Carcinoma
Brief Title: PD-1 Inhibitor Combined With Neoadjuvant Chemotherapy in Subjects With Resectable Locally Advanced Thoracic Esophageal Squamous Cell Carcinoma
Acronym: REVO
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fujian Cancer Hospital (Other Government)
Collaborators: Suzhou Suncadia Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OBU-FJ-EC-II-007
Record Dates: First submitted 2021-08-10; First posted 2021-08-16 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-11

CONDITIONS: Esophageal Neoplasms; Esophageal Squamous Cell Carcinoma
Keywords: Neoadjuvant; Esophageal Cancer; PD-1 Inhibitor
MeSH Terms: conditions — Esophageal Neoplasms; Esophageal Squamous Cell Carcinoma | interventions — Immune Checkpoint Inhibitors; Albumin-Bound Paclitaxel; Cisplatin; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PD-1 Inhibitor+albumin-bound paclitaxel+cisplatin (Experimental): Participants receive PD-1 Inhibitor 200mg on Day 1 every 3 weeks (Q3W), albumin-bound paclitaxel 125 mg/m^2 on Day 1, 8 Q3W, and cisplatin 75 mg/m^2 on Day 1 Q3W, a total of 2-4 cycles，followed by surgery.
  Interventions: Drug: PD-1 inhibitor; Drug: Albumin-Bound Paclitaxel; Drug: Cisplatin
- Albumin-bound paclitaxel+cisplatin+radiotherapy (Active Comparator): Participants receive albumin-bound paclitaxel 125 mg/m^2 on Day 1, 8 Q3W, and cisplatin 75 mg/m^2 on Day 1 Q3W, a total of 2 cycles combined with radiotherapy(40Gy/2Gy),followed by surgery.
  Interventions: Drug: Albumin-Bound Paclitaxel; Drug: Cisplatin; Radiation: Radiation

INTERVENTIONS:
Drug: PD-1 inhibitor — PD-1 Inhibitor 200mg D1 Q3W
  Arms: PD-1 Inhibitor+albumin-bound paclitaxel+cisplatin
Drug: Albumin-Bound Paclitaxel — 125 mg/m^2 D1/D8 Q3W
Drug: Cisplatin — 75 mg/m^2 D1 Q3W
Radiation: Radiation — 40Gy/2.0Gy
  Arms: Albumin-bound paclitaxel+cisplatin+radiotherapy

SUMMARY:
The purpose of this study is to explore the efficacy and safety of compare the efficacy and safety of PD-1 inhibitor and chemotherapy（treatment group） with chemoradiotherapy（control group） in neoadjuvant treatment of resectable thoracic esophageal squamous cell carcinoma.

DETAILED DESCRIPTION:
This is a randomized, open-label, phase II study of PD-1 inhibitor combined With neoadjuvant chemotherapy versus neoadjuvant chemoradiotherapy in subjects With resectable locally advanced thoracic esophageal squamous cell carcinoma. The patients will be divided into two groups(1:1). In the treatment group, PD-1 inhibitor ,albumin-bound paclitaxel and cisplatin will be given every 3 weeks for 2-4 cycles as neoadjuvant therapy. In the control gourp, albumin-bound paclitaxel and cisplatin will be given every 3 weeks for 2 cycles as neoadjuvant therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteered to participate in the study, signed the informed consent form;
2. Histologically or cytological confirmed esophageal squamous cell carcinoma;
3. Patients with resectable disease of primary tumor in thoracic esophagus (cT1b-4aN1-3M0, cT3-4aN0M0) evaluated by CT/MRI/EUS;
4. Expected R0 resection;
5. Aged 18-75 years, male or female;
6. ECOG PS 0-1;
7. Without prior treatments including surgery, chemotherapy, radiotherapy, and targeting treatment for esophageal cancer;
8. Surgery is planned after neoadjuvant treatment;
9. Without any contraindication of operation;
10. Adequate organ function as follows: 1) Routine blood test: Leukocytes >=3.0x10^9/L; Absolute neutrophil count >=1.0x10^9/L; Platelet >=80x10^9/L; Hemoglobin >=90 g/L; 2) Blood biochemical test: Total bilirubin <=1.5 ULN; ALT <=2.5 ULN; AST <=2.5 ULN; Serum creatinine <=1.5 ULN or creatinine clearance rate >=50 mL/min (Cocheroft-Gault); 3) Coagulation function test: INR <=1.5 ULN; APTT <=1.5 ULN;
11. For females of child bearing potential, a negative serum/urine pregnancy test result within 72h before study treatment. For female and male participants of reproductive potential must be willing to use adequate contraception for the course of the study until 3 months after the last dose of any of the drugs in the study;
12. Had good compliance and cooperated with the follow-up.

Exclusion Criteria:

1. The tumor invades the adjacent organs of the esophageal lesion (aorta or trachea);
2. Patients with supraclavicular lymph node metastasis;
3. Uncontrollable pleural effusion, pericardial effusion or ascites requiring repeated drainage;
4. Poor nutritional status, BMI < 18.5 Kg/m2; If corrected after nutritional support before randomization, enrollment can be further considered after evaluation by the principal investigator;
5. Has a history of allergy to monoclonal antibody, any component of PD-1 Inhibitor, paclitaxel, cisplatin or other platinum drugs;
6. Has received or is receiving any of the following treatments: A)any anti-tumor radiation, chemotherapy or other treatment drugs; B) Immunosuppressive drugs or whole-body hormone drugs are being used for immunosuppressive purposes within 2 weeks prior to the first use of the study drug (dose > 10mg/ day prednisone or equivalent dose);Inhalation or topical use of steroids and 10 mg/ day prednisone or equivalent dose of adrenocortical hormone replacement is permitted in the absence of active autoimmune disease; C) Received attenuated vaccine within 4 weeks before the first use of the study drug; D) Major surgery or severe trauma within 4 weeks prior to the first use of the study drug;
7. History of any active autoimmune disease, including but not limited to: interstitial pneumonia, enteritis, hepatitis, hypohysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism (may be considered after hormone replacement therapy);Patients with psoriasis or childhood asthma/allergy who have been in complete remission and do not need any intervention as adults may be considered for inclusion, but patients requiring medical intervention with bronchodilators may not be included;
8. History of immunodeficiency, including HIV positive, or other acquired or congenital immunodeficiency disease, or history of organ transplantation or allogeneic bone marrow transplantation;
9. Present of poorly controlled cardiac symptoms or disease, including but not limited to: (1) heart failure with NYHA class II or above (2) unstable angina, （3）myocardial infarction occurred within 1 year (4) clinical significance supraventricular or ventricular arrhythmias without clinical intervention or poorly controlled after clinical intervention;
10. Severe infection (CTCAE > 2) occurred within 4 weeks prior to the first use of the study drug, such as severe pneumonia, bacteremia, infection complications requiring hospitalization, etc.;Baseline chest imaging indicated active pulmonary inflammation, infection signs and symptoms within 14 days prior to the first use of the study drug, or the need for oral or intravenous antibiotic treatment, except prophylactic antibiotic usage;
11. Patients who are found to have active pulmonary tuberculosis infection through medical history or CT, or have active pulmonary tuberculosis infection history within 1 year before enrollment, or have active pulmonary tuberculosis infection history more than 1 year before but without regular treatment;
12. Have hereditary bleeding tendency or coagulation dysfunction. There were clinically significant bleeding symptoms or a clear bleeding tendency within 3 months before enrollment, such as gastrointestinal bleeding, hemorrhagic gastric ulcer, fecal occult blood++ and above at baseline;
13. Active hepatitis B (HBV DNA ≥ 2000 IU/mL or 10^4 copies/mL), hepatitis C (HCV antibody positive, and HCV RNA higher than the detection limit of analytical method);
14. Other malignancies diagnosed within 5 years prior to the first use of the study drug, except those with a low risk of metastasis or death (5-year survival rate > 90%), such as adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix;
15. Pregnant or lactating women;
16. In the investigator's judgment, there were other factors that might have contributed to the forced termination of the study, such as the need for combined treatment with other serious medical conditions (including mental illness), alcohol and drug abuse, family or social factors that might have affected the safety or compliance of the subjects.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2021-08-15 (Actual); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Pathologic complete response (pCR) rate | Within 14 working days after surgery

SECONDARY OUTCOMES:
R0 resection rate | Within 14 working days after surgery
Overall Survival (OS) | Up to 8 years
  OS is defined as the time from randomization until death from any cause.
Disease Free Survival (DFS) | Up to 8 years
  The time from the first day of the date of surgery to local or distant recurrence, or death caused by any cause, whichever occurs first;

CONTACTS AND LOCATIONS:
Overall Officials: Shuoyan Liu, Study Chair — Fujian Cancer Hospital
Locations (6):
- China (6):
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - the Second Hospital of Longyan, Longyan, Fujian
  - the First Hospital of Putian City, Putian, Fujian
  - Fujian Medical University 2nd Affiliated Hospital, Quanzhou, Fujian
  - Quanzhou First Hospital, Quanzhou, Fujian
  - the First Affiliated Hospital of Xiamen University, Xiamen, Fujian